CLINICAL TRIAL: NCT03351491
Title: Use of Smartphone Health Applications Among Patients Aged 18 to 69 Years Recruited in Primary Care in Grenoble Area
Acronym: Smartcheck
Status: Completed | Type: Observational
Sponsor: University Grenoble Alps (Other)
Responsible Party: Principal Investigator, Roussel Jérémy, Principal Investigator, University Grenoble Alps
Other Study IDs: 2017-A01647-46
Record Dates: First submitted 2017-11-08; First posted 2017-11-22 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Mobile Applications; Mobile Health
Keywords: Health mobile applications; Apps; mhealth; ehealth; France; msanté; applications mobiles

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the frequency of use of smartphone health applications among people consulting in primary care in the Grenoble region, France.

This is a descriptive study using a questionnaire completed by the patient and distributed by general practitioners. The study also collects the type of used application as well as the rhythm of usage, and compares the use of mobile health applications according to the sociodemographic, geographical and medical characteristics of the studied population.

DETAILED DESCRIPTION:
Smartphones are more and more present and change many aspects of people's life, especially in the field of health. The appearance of numerous mobile health applications over the past years explains this strong attractiveness.

According to some studies, these could lead to savings in health care systems by promoting a preventive approach and refocusing cares on the patient who would be more independent. However, not much data on the use of smartphone health applications by patients are reported in the scientific literature.

The main objective of this study is to evaluate the frequency of use of smartphone mobile health applications among primary care patients aged 18 to 69 in the Grenoble region, France.

The secondary objectives are the collection of the kind of application used, the rhythm of usage of these health applications and the comparison of the frequency of use with the sociodemographic, geographical and medical characteristics of the studied population.

To this end, the investigators use a questionnaire distributed by voluntary general practitioners and filled by patients. The number of subjects to be included is 385 and the number of distributed questionnaires is 1500.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged among 18 to 69 years old who consults a general practitioner regardless of the reason for consultation

Exclusion Criteria:

* patients aged 17 and less and patients aged 70 years and over.
* Patients not owning a mobile phone and / or smartphone for own
* Patients deprived of their liberty by judicial or administrative decision or subject to a legal protection measure

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population recruited in 12 general practictioners and 1 primary care center in Grenoble area in France.
Sampling Method: Non-Probability Sample
Enrollment: 597 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-01-07 (Actual); Study Completion 2018-01-14 (Actual)

PRIMARY OUTCOMES:
Use of at least one mobile health application on a smartphone | month 1
  Use of at least one mobile health application on a smartphone since the first use of a smartphone.

SECONDARY OUTCOMES:
Socio-demographic characteristics | month 1
  Age (years) Sex (F/M) socio-professional group
Geographical characteristics | month 1
  Postcode
Names of applications used by the patient | month 1
  The patient name the applications which he used. In order to help him/her , there are some examples of kind of applications.
Origin of the awareness of the existence of the mobile health application used. | month 1
  How the patient became aware of the existence of used application: general practitioners, other doctors, other health professionals, media, social circle
Number of drugs on the prescription | month 1
  number of drugs on the prescription.
Illness requiring treatment for more than a year | month 1
  Diabetes, malignant tumor, psychiatric condition, cardiac diseases, rheumatological diseases, pulmonary diseases, chronic renal failure, other

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - Dr Ronflet, Châbons
  - Centre de santé de l'abbaye, Grenoble
  - Dr CROS, Grenoble
  - Dr Grasset, Grenoble
  - Dr Riehl, La Côte-Saint-André
  - Dr Fuentes, Meylan
  - Maison médicale Moirans, Moirans
  - Dr PARADIS, Montmélian
  - Dr Chatellard, Saint-Martin-d'Hères
  - Dr Moulis, Saint-Martin-d'Hères
  - Maison médicale Saint Martin d'Hères, Saint-Martin-d'Hères
  - Maison Médicale de Tullins, Tullins
  - Dr Bichon, Villard-de-Lans

REFERENCES:
- [Derived] Paradis S, Roussel J, Bosson JL, Kern JB. Use of Smartphone Health Apps Among Patients Aged 18 to 69 Years in Primary Care: Population-Based Cross-sectional Survey. JMIR Form Res. 2022 Jun 16;6(6):e34882. doi: 10.2196/34882. PMID 35708744